CLINICAL TRIAL: NCT00825071
Title: Optimizing Anesthesia Antiemetic Measures Versus Combination With Dexamethasone or Ondansetron in the Prevention of Postoperative Nausea and Vomiting.
Brief Title: Dexamethasone for Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Subhi M. Alghanem, Professor of Anesthesia and Intensive Care, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UJordan
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Ondansetron; Dexamethasone
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone; Ondansetron; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group D (Active Comparator): Dexamethasone group : This group received 8 mg dexamethasone
  Interventions: Drug: Dexamethasone
- Group O (Active Comparator): Ondansetron Group: received 4 mg ondansetron
  Interventions: Drug: Ondansetron
- Group P (Placebo Comparator): (Group P) received normal saline (Placebo)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Dexamethasone — 8 mg, Intravenous
  Arms: Group D
Drug: Ondansetron — 4 mg, intravenously
  Arms: Group O
Drug: normal saline — 2 ml, intravenously
  Arms: Group P

SUMMARY:
The investigators want to test the efficacy of these anesthetic antiemetic measures collectively with or without ondansetron or dexamethasone, in the prevention of postoperative nausea and vomiting (PONV) in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
More than half of the patients undergoing laparoscopic cholecystectomy will have postoperative nausea and vomiting (PONV). PONV is related to surgical, anesthetic and patient factors.

We want to test the efficacy of these anesthetic antiemetic measures collectively with or without ondansetron or dexamethasone, in the prevention of PONV in patients undergoing laparoscopic cholecystectomy.

Three groups to be studied : (Group O) will receive 4 mg ondansetron, (Group D) will receive 8 mg dexamethasone and (Group P) will receive normal saline .

ELIGIBILITY:
Inclusion Criteria:

* (ASA) grade I and II, aged (18-70 years) who are scheduled for elective laparoscopic cholecystectomy under general anesthesia at the department of Anesthesia and Intensive Care, University of Jordan, Amman, Jordan between November 2007 and March 2008

Exclusion Criteria:

* All patients who received antiemetics or cortisone within 48 hr before surgery or those who required opioids before and after surgeries
* Pregnant, breast feeding ladies
* Any patient with BMI (Body Mass Index) > 34 kg/m²
* Patient with gastrointestinal, hepatic, renal, mental or psychiatric illnesses or those with history of motion sickness were also excluded from the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
incidence of nausea and vomiting in each of the three studied groups. | 5 months

SECONDARY OUTCOMES:
Assess the postoperative Visual Analog Score for pain assessment in each of the three studied groups | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Subhi M Al-Ghanem, MD, FFARCSI, Principal Investigator — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Background] Macario A, Weinger M, Carney S, Kim A. Which clinical anesthesia outcomes are important to avoid? The perspective of patients. Anesth Analg. 1999 Sep;89(3):652-8. doi: 10.1097/00000539-199909000-00022. PMID 10475299
- [Result] Watcha MF, White PF. Postoperative nausea and vomiting. Its etiology, treatment, and prevention. Anesthesiology. 1992 Jul;77(1):162-84. doi: 10.1097/00000542-199207000-00023. PMID 1609990
- [Result] Thune A, Appelgren L, Haglind E. Prevention of postoperative nausea and vomiting after laparoscopic cholecystectomy. A prospective randomized study of metoclopramide and transdermal hyoscine. Eur J Surg. 1995 Apr;161(4):265-8. PMID 7612769
- [Result] Apfel CC, Kranke P, Katz MH, Goepfert C, Papenfuss T, Rauch S, Heineck R, Greim CA, Roewer N. Volatile anaesthetics may be the main cause of early but not delayed postoperative vomiting: a randomized controlled trial of factorial design. Br J Anaesth. 2002 May;88(5):659-68. doi: 10.1093/bja/88.5.659. PMID 12067003
- [Result] Nesek-Adam V, Grizelj-Stojcic E, Rasic Z, Cala Z, Mrsic V, Smiljanic A. Comparison of dexamethasone, metoclopramide, and their combination in the prevention of postoperative nausea and vomiting after laparoscopic cholecystectomy. Surg Endosc. 2007 Apr;21(4):607-12. doi: 10.1007/s00464-006-9122-7. Epub 2007 Feb 7. PMID 17285386
- [Result] Chohedri AH, Matin M, Khosravi A. The impact of operative fluids on the prevention of postoperative anesthetic complications in ambulatory surgery--high dose vs low dose. Middle East J Anaesthesiol. 2006 Oct;18(6):1147-56. PMID 17263269
- [Result] Cechetto DF, Diab T, Gibson CJ, Gelb AW. The effects of propofol in the area postrema of rats. Anesth Analg. 2001 Apr;92(4):934-42. doi: 10.1097/00000539-200104000-00027. PMID 11273930
- [Result] Tramer MR, Reynolds DJ, Moore RA, McQuay HJ. Efficacy, dose-response, and safety of ondansetron in prevention of postoperative nausea and vomiting: a quantitative systematic review of randomized placebo-controlled trials. Anesthesiology. 1997 Dec;87(6):1277-89. doi: 10.1097/00000542-199712000-00004. PMID 9416710